CLINICAL TRIAL: NCT06513715
Title: Discovery of Bioactive Compounds as Agonists of GLP1 Receptor for Obesity Treatment
Brief Title: Activity of Bioactive Natural Compounds as Potential Agonists of GLP1R
Acronym: BIOBESICOM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Juan Jose Hernández Morante, Faculty of Nursing Research Coordinator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIOBESICOM
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Obesity; Overweight
Keywords: weight loss; prickly pear; obesity; overweight; appetite; hunger; satiety
MeSH Terms: conditions — Obesity; Overweight; Weight Loss | interventions — jubanine C

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CONTROL (Placebo Comparator): The participants allocated in this arm will follow a treatment with placebo
  Interventions: Dietary Supplement: Control
- Intervention 1 (Experimental): The participants in this arm will receive a 150 mg dose of jubenine
  Interventions: Dietary Supplement: Jubanine
- Intervention 2 (Experimental): The participants in this arm will receive a 300 mg dose of jubenine
  Interventions: Dietary Supplement: Jubanine
- Intervention 3 (Experimental): The participants in this arm will receive a 300 mg dose of prickly pear extract
  Interventions: Dietary Supplement: Jubanine

INTERVENTIONS:
Dietary Supplement: Control — This intervention will be made with a placebo
  Arms: CONTROL
Dietary Supplement: Jubanine — This intervention will be made with jubanine or prickly pear extract
  Arms: Intervention 1; Intervention 2; Intervention 3

SUMMARY:
The goal of this clinical trial is to learn if natural bioactive compound jubenine works to reduce appetite and to favour weight loss. It will also learn about the safety of natural bioactive compound jubenine. The main questions it aims to answer are:

Does natural bioactive compound jubenine reduce the hunger perception or increase the satiety perception, and, consequently, reduce food intake? What medical problems do participants have when taking natural bioactive compound jubenine? Researchers will compare natural bioactive compound jubenine to a placebo (a look-alike substance that contains no drug) to see if natural bioactive compound jubenine works to reduce food intake for obesity treatment.

Participants will:

Take natural bioactive compound jubenine or a placebo three times every day for 3 months.

Visit the clinic once every 1 week for checkups and tests. Keep a diary of their symptoms and potenital adverse effects.

DETAILED DESCRIPTION:
The general objective of the present project is to confirm the activity of non-peptide compounds from bioactive natural sources, concretely jubenine, which will be a GLP1R agonists for their potential therapeutic usefulness for the treatment of obesity.

The objective of the present trial was the determination of the effectiveness for weight loss, through a preclinical trial, of those compounds with the greatest potential, which according to our previous data, is jubenin.

The design of the present study is a double-blind, randomized, placebo-controlled, crossover pilot trial conducted on healthy men and women volunteers. Individuals will be randomized to receive placebo, one of a range of jubenine doses, and a nopal extract for 7 days, where participants will be maintained on a precisely controlled diet along the different interventions. Each subject will receive three standardized meals daily with 30% of calories from fat. On the intervention days, meals will be distributed at breakfast, lunch and dinner, along with one of the indicated doses according to their randomization. Meals were distributed at 08:30, 13:30 and 20:00, trying to adjust to the patients' habits. A nurse will be present during the distribution of meals to ensure the intake of the compound.

All treatments will be delivered on green capsules, size 0, made with hard gelatin (head and body) (provided by Guinama Ltd, Valencia, Spain). These capsules are capable of disintegrating in less than 15 minutes and meet the requirements of the European Pharmacopoeia and USP. Capsucel (microcrystalline cellulose, Guinama Ltd, Valencia, Spain), will be employed as excipient in all treatments. Jubenine will be extracted from prickly pears following standard chemistry procedures. Jubenine, a prickly pear extract, with a 50% of jubanine content, will be obtained from Metapharmaceuticals (Metapharmaceuticals Ltd, Barcelona, Spain). The treatments will be made by two researchers, who will not be present at the time of administration. These researchers will also carry out the randomization, according to a Latin Square procedure, to ensure that all participants followed all the interventions. Randomization will be performed by a member of the research group with Excel software, with a visual basic Macro developed to this end.

Each study will comprise an initial screening visit one week prior to the start of the study, with a 1-day run-in period, 7-day treatment period and a 1-day post-treatment follow-up visit. The initial evaluation will be carried out by a physician, where a complete physical examination will be performed. This will allow us to exclude the presence of any disease or disorder in the participants, so all volunteers took part in the study.

The main endpoint of the effectiveness of the study will be changes in hunger/satiety sensations, determined by a visual analogic scale. Secondary endpoints will be clinical signs, and tolerability (gastrointestinal adverse effects), and clinical laboratory parameters, in particular, cholesterol, high-density lipoprotein (HDL-C), low-density lipoprotein (LDL-C), and triglycerides.

ELIGIBILITY:
Inclusion Criteria:

* BMI over 24.9
* no clinically relevant abnormalities and no relevant systemic disease history

Exclusion Criteria:

* the presence of any clinically relevant symptoms or severe disease within 4 weeks of the start of the study
* any history of hepatic dysfunction, any condition that might affect the pharmacokinetics properties of the study drug.
* diarrhoea (>2 liquid stools per day) or constipation (3 days duration) 1 week prior to the start of the study
* history of hypersensitivity to GLP1R agonists
* evidence of hepatitis B or C, HIV positivity
* smoking (>4 cigarettes/day)
* history of alcohol or substance abuse
* bulimia or laxative abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Weight loss | First evaluation will be made after 3 months of treatment, and a second evaluation will be made 12 months later.
  Percentage of weight loss from baseline weight

CONTACTS AND LOCATIONS:
Overall Officials: Juan José Hernández Morante, PhD, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (1):
- Faculty of Nursing. Catholic University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available after ending the study.
Access Criteria: Study protocol and statistical plan will be available online for all users. Informed consent form and clinical study report will be accesible under reasonable request.